CLINICAL TRIAL: NCT06721351
Title: Diabetic Retinopathy Screening Point-of-Care Artificial Intelligence -DRES-POCAI: AI - Clinical Intervention at San Ysidro Health
Brief Title: Diabetic Retinopathy Screening Point-of-Care Artificial Intelligence
Acronym: DRES POCAI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro De Salud La Comunidad De San Ysidro Inc DBA: San Ysidro Health (Other)
Collaborators: Eyenuk, Inc. (Industry); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Fatima Muñoz, Associate Vice President Health Support Services, Centro De Salud La Comunidad De San Ysidro Inc DBA: San Ysidro Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RHP-091323-159; 212825-SYH-04 (Other: Kaiser Permanente)
Record Dates: First submitted 2024-11-20; First posted 2024-12-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Retinopathy (DR)
Keywords: Point-of-care (POC) artificial intelligence (AI) technology for DR screening; Diabetic Retinopathy (DR) Screening; Diabetes
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The DRES-POCAI study uses a randomized controlled, open-label, parallel superiority trial.
  Randomization: Participants will be randomized into two groups: usual care (receive a retinal screening by an optometrist) or intervention group (receive a retinal screening using a special camera and FDA-cleared EyeArt® system, an autonomous AI-based DR screening).
  Open-label Design: Blinding participants and providers to the autonomous DR screening is logistically difficult. The intervention's immediate results and potential impact on the workflow necessitate an open-label approach.
  Parallel Design: The parallel design allows for a clear, side-by-side comparison of outcomes between the intervention and usual care groups over time.
  Superiority Evaluation: The primary objective is to determine if the multi-component DRES-POCAI intervention is superior to usual care in increasing DR screenings, early detection, referrals, and patient knowledge/self-efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Usual care (No Intervention): The usual care group will complete the DR screening with an eye care provider on a different day and at a different location. The study staff will facilitate this process for participants in the usual care group by assisting them in scheduling appointments for their routine retinal screening.
- Diabetic Retinopathy Screening (Experimental): The intervention group will complete the DR screening using a special camera and the AI system (EyeArt®), the same day of the study visit. Participants assigned to the intervention group will also receive a retinal screening without dilation using the EyeArt® AI system; the DR screening will be completed before their medical provider visits. The results will be available immediately after the screening, allowing participants to learn about and discuss their eye health with their care provider.
  Interventions: Diagnostic Test: Diabetic Retinopathy screening Point of Care Artificial Intelligence

INTERVENTIONS:
Diagnostic Test: Diabetic Retinopathy screening Point of Care Artificial Intelligence — Random assignment of participants to intervention and control groups minimizes confounding variables. This ensures that any observed differences in outcomes are likely due to the intervention itself and not pre-existing differences between the groups. Participants of the DRES-POCAI study will be randomized into two groups: usual care (receive a retinal screening by an optometrist) or intervention group (receive a retinal screening using a special camera and EyeArt® system, an autonomous AI-based DR screening). The randomization will occur after consenting and completing the surveys, prior to conducting the DR screening process (for those randomized to the intervention group).
  Arms: Diabetic Retinopathy Screening

SUMMARY:
This research study is being conducted to improve eye care by using artificial intelligence (AI) to make diabetic eye screenings faster and more accessible. AI technology mimics human decision-making, enabling computers and systems to analyze medication information. Specifically for this screening, AI examines digital images of the eye and based on that information, may identify if a participant has diabetic retinopathy. It can assist doctors in making decisions about a participant's diagnosis, treatment or care plans to improve patient care. This is a collaboration between San Ysidro Health (SYHealth), University of California, San Diego (UC San Diego), and Eyenuk. The Kaiser Permanente Augmented Intelligence in Medicine and Healthcare Initiative (AIM-HI) awarded SYHealth funds to demonstrate the value of AI technologies in diverse, real-world settings.

DETAILED DESCRIPTION:
This study is intended to address unmet medical needs in diabetic eye care in a community health center setting by enhancing and modifying existing clinical practices with the integration of point-of-care (POC) artificial intelligence (AI) technology for Diabetic Retinopathy (DR) screening. Using a special camera and a computer system called EyeArt® to make diabetic eye screenings faster and more accessible. EyeArt®, is a Food Drug and Administration (FDA)-cleared device system for fast, non-invasive Diabetic retinopathy screening. This non-invasive DR screening does not require dilation and provides immediate results and facilitates informed discussions with their primary care provider. This study will optimize, implement, and test the impact of a multicomponent intervention that includes: 1) autonomous DR screening, a fast and non-invasive retinal exam into the primary care settings with 2) integration of the results into the EHR and 3) health education/care coordination support (e.g., patient education). Primary Objective (Clinical): Evaluate the implementation and effectiveness of a multicomponent AI clinical intervention on DR screenings rate, early stages of DR detection, and referrals to the specialist for follow up on abnormal results. Secondary Objectives: Evaluate the implementation and effectiveness of a multicomponent AI clinical intervention on DR knowledge, attitudes, self-efficacy, and patient satisfaction.

Participants will be active SYHealth patients 22 years of age or older with diabetes mellitus (DM) who have not had a retinal exam in the last 11 months, and have a medical visit scheduled during the intervention period and are able to read and understand either English or Spanish in order to provide informed consent and complete study surveys. Exclusion criteria: 1) have a prior diagnosis of DR, macular edema, or retinal vascular occlusion; 2) have persistent visual Impairment in one or both eyes; 3) history of ocular injections, laser treatment of the retina, or intraocular surgery (excluding cataract surgery); 4) pregnant women; and 5) diagnosis of mental or degenerative disease that prevents self-consent for the study. The study will recruit a cohort of 848 adults from two SYHealth clinic sites.

Once the potential participants arrive at their study visit appointment, they will complete the consent process, pre-survey (knowledge, attitudes and self-efficacy about diabetes and eye health). Participants will be randomized into either the DR screening-AI-intervention or retinal screening usual care groups and continue study activities as follows:

1. Participants assigned to the DR screening-AI-intervention group will undergo DR screening in-clinic prior to the medical visit using a special camera and the EyeArt® Artificial Intelligence (AI) system (Eyenuk, Inc.), an FDA-cleared AI device for fast, non-invasive DR screening. This screening, which does not require dilation, uses a camera with a smart computer technology using AI that can detect signs of significant diabetic retinopathy in less than five minutes. These results will be immediately integrated into the electronic health record (EHR), enabling informed discussions with their primary care provider at the time of their medical visit and will automatically generate the referrals to an eye specialist for participants with abnormal findings. Participants will receive a copy of the results immediately after completion of the screening. After the screening, participants will receive a copy of the results of the screening, health education information on DR and eye health before completing their baseline study visit. Subsequently, they will proceed with their medical visit to ensure continuity of their diabetes care.
2. Participants in the retinal screening usual care group will receive assistance from the RA to schedule the appointment with an eye care provider according to SYHealth's protocols for routine retinal screening, which includes dilation. After the RA scheduled the visit with the eye care provider, participants will receive health education information on DR and eye health before completing their baseline study visit. Subsequently, they will proceed with their medical visit to ensure continuity of their diabetes care.

Appointments with the eye care provider are usually at a different clinic location based on availability, and the retinal screenings are not completed on the same day of the medical visit with their primary care provider. At the time of the visit with the eye care provider will discuss the retinal screening results with the participant and may conduct a comprehensive eye exam, submitting referrals for any abnormal results.

ELIGIBILITY:
Inclusion Criteria:

1. Capacity to provide informed consent. Individuals must have the capacity to understand the study information, risks, and benefits and voluntarily provide informed consent.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Established and active patient of SYHealth-CV and KC (having a medical appointment in the last 18 months).
4. Person aged 22 and older.
5. Established diagnosis of DM.
6. Medical appointment(s) (in-person or telehealth) scheduled during the intervention period.
7. Has not completed a dilated eye exam or retinal exam in the last 11months.

Exclusion Criteria:

1. have a prior diagnosis of DR, macular edema, or retinal vascular occlusion;
2. have persistent visual Impairment in one or both eyes;
3. history of ocular injections, laser treatment of the retina, or intraocular surgery (excluding cataract surgery);
4. pregnant women; and
5. diagnosis of mental or degenerative disease that prevents self-consent for the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2024-07-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
DR screening completion and result | the enrollment (baseline) and through study completion, an average of 1 year
  1. Completion of DR screening. Data obtained through EHR at the time of the enrollment (baseline) and through study completion, an average of 1 year.
  2. Results of DR screening: usual care specific diagnosis; intervention group defined as normal, mild-to-moderate DR), visual threatening DR or ungradable. Referral to specialist completion status and final diagnosis.
DR screening efficiency | the enrollment (baseline) and through study completion, an average of 1 year
  EyeArt system impact and efficiency data, number of orders submitted, screenings completed (images), number of ungradable and time of attempts, time (minutes) the participant spent in front of the camera.
Knowledge and attitudes about DR | Baseline survey at study visit and follow up survey 6-months after.
  5 min-survey at baseline and 6 months. Assessment of participant knowledge and attitudes about DR (10 multiple choice question survey).
DM self-efficacy | Baseline survey at study visit and follow up survey 6-months after.
  5 min-survey at baseline and 6 months. Assessment of participant DM self-efficacy (seven questions using a 5-point scale from "Strongly disagree" to "Strongly agree).
DM self-management | Baseline survey at study visit and follow up survey 6-months after.
  5 min-survey at baseline and 6 months. Assessment of participant DM self-management ( 5-point scale from "Very difficult: I couldn't do it at all" to "Not difficult: I could do all of I).
DR Screening Satisfaction Survey (Intervention Group) | Baseline survey at study visit and follow up survey 12-months after (at next DR screening).
  5 min-survey at baseline and 6 months. Assessment of participant satisfaction with POC DR screening (three questions using a 5-point scale from "Strongly disagree" to "Strongly agree, three multiple choice questions, and one open text field).
Demographic and Clinical Data | Intake at study 1 day visit.
  Participant level demographics (e.g., sex assigned at birth, gender, age, race, ethnicity, marital status, employment status, insurance type etc.) and clinical data will be extracted from the electronic health record to obtain participant level information on comorbidities, medication use and compliance with quality methods and as applicable selected patient visit history.
Social Determinants of Health | Intake at study 1 day visit.
  Participant information on non-medical factors (e.g., socioeconomic status, employment, housing stability, food insecurity, education, social support networks, living environment, alcohol/tobacco consumption) that could influence health outcomes will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Muñoz, MD, MPH, Principal Investigator — San Ysidro Health; Nicole Stadnick, PhD, Principal Investigator — University of California, San Diego
Locations (3):
- United States (3):
  - San Ysidro Health Chula Vista, Chula Vista, California
  - San Ysidro Health - Comprehensive Health Center - Ocean View, San Diego, California
  - San Ysidro Health King-Chavez Health Center, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diaz EA, Seifert ML, Gruning V, Stadnick NA, Lugo-Butler E, Servin AN, Rodriguez-Rosales CI, Geremia C, Ramachandra C, Bhaskaranand M, Howard D, Solis O, Velasquez S, Snook B, Tucker S, Munoz FA. Diabetic Retinopathy Screening Among Federally Qualified Health Center Patients Using Point-of-Care AI: DRES-POCAI: A Trial Protocol. JAMA Netw Open. 2025 Oct 1;8(10):e2538114. doi: 10.1001/jamanetworkopen.2025.38114. PMID 41118165